CLINICAL TRIAL: NCT01534078
Title: Brentuximab Vedotin Plus AVD in Non-bulky Limited Stage Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin Plus AVD in Limited-stage Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Seagen Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-462
Record Dates: First submitted 2012-02-09; First posted 2012-02-16 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Hodgkin Lymphoma
Keywords: non-bulky; limited stage
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Brentuximab Vedotin in combination with Adriamycin, Vinblastine and Dacarbazine
  Interventions: Drug: Brentuximab Vedotin; Drug: Adriamycin, vinblastine, and dacarbazine

INTERVENTIONS:
Drug: Brentuximab Vedotin — 2 doses administered 14 days apart; followed by combination therapy with AVD for 4-6 cycles; 1.2 mg/kg
  Other Names: Adcetris; SGN-35; SGN35
Drug: Adriamycin, vinblastine, and dacarbazine — Combination therapy with brentuximab for 4-6 cycles; 25 mg/m2 Adriamycin; 6 mg/m2 Vinblastine; 375 mg/m2 Dacarbazine
  Other Names: Doxorubicin; Velban; DTIC

SUMMARY:
Brentuximab is an antibody-drug conjugate (ADC), which is the combination of an antibody (a protein that binds to cells) and a chemotherapy molecule. Brentuximab works by using the antibody portion to enter into the Hodgkin lymphoma cells and then releasing the chemotherapy portion, which attempts to destroy the cell.

The intravenous chemotherapy drugs Adriamycin, Vinblastine and Dacarbazine (AVD) which you will receive in this research study are approved for use in people with Hodgkin Lymphoma. A drug called bleomycin is usually included with AVD, but since it appears to be a less effective drug with significant potential risks, it is being replaced in this study with the drug brentuximab.

In this research study, the investigators are looking to see whether brentuximab in combination with AVD is effective in treating limited-stage Hodgkin Lymphoma.

DETAILED DESCRIPTION:
Each treatment cycle is 28 days. You will receive brentuximab alone on Day 1 and 15 of the first cycle (lead-in cycle). After cycle 1, you will receive brentuximab combined with AVD on Day 1 and 15 for 4-6 cycles, depending on your response to therapy. Brentuximab and AVD will be given to you by intravenous infusion (IV).

The following test and procedures will be performed on Days 1 and 15 of each cycle:

* Review of any side effects you have experienced and all medications you are taking
* Performance Status
* Physical exam and vital signs
* Routine blood tests
* Questionnaire to evaluate symptoms of neuropathy
* Research blood sample to look at markers to see how your body is responding to study medication
* PET-CT scan prior to completing cycle 2 of combination brentuximab/AVD

After the final dose of the study drug: The following assessments will be performed within one month of your last dose of study medication:

* Review of any side effects you have experienced and all medications you are taking
* Performance Status
* Physical exam and vital signs
* Routine blood tests
* Questionnaire to evaluate symptoms of neuropathy
* Research blood sample to look at markers to see how your body is responding to study medication
* PET-CT scan Follow up will include the following
* Review of any side effects you have experienced and all medications you are taking
* Performance Status
* Review and Physical exam
* Routine blood tests
* Questionnaire to evaluate symptoms of neuropathy
* CT scans

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated stage IA, IB, IIA or IIB classical Hodgkin Lymphoma
* Non-bulky disease defined as less than 10 cm in maximal diameter
* Measurable disease greater than or equal to 1.5 cm
* ECOG performance status of 0 or 2
* Willing to use 2 effective forms of birth control

Exclusion Criteria:

* No prior chemotherapy or radiotherapy for Hodgkin lymphoma
* Not receiving any other investigational agents
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to Adriamycin, Vinblastine, Dacarbazine or brentuximab
* No pre-existing grade 3 or greater neuropathy
* No uncontrolled intercurrent illness
* Not pregnant or breastfeeding
* No history of a different malignancy unless disease free for at least one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, M.D., Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Abramson JS, Arnason JE, LaCasce AS, Redd R, Barnes JA, Sokol L, Joyce R, Avigan D, Neuberg D, Takvorian RW, Hochberg EP, Bello CM. Brentuximab vedotin, doxorubicin, vinblastine, and dacarbazine for nonbulky limited-stage classical Hodgkin lymphoma. Blood. 2019 Aug 15;134(7):606-613. doi: 10.1182/blood.2019001272. Epub 2019 Jun 11. PMID 31186274

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Brentuximab Vedotin in combination with Adriamycin, Vinblastine and Dacarbazine (AVD)
  Brentuximab Vedotin: 2 doses administered 14 days apart; followed by combination therapy with AVD for 4-6 cycles; 1.2 mg/kg
  Adriamycin, vinblastine, and dacarbazine: Combination therapy with brentuximab for 4-6 cycles; 25 mg/m2 Adriamycin; 6 mg/m2 Vinblastine; 375 mg/m2 Dacarbazine
Period: Overall Study
Arm/Group | Treatment Arm
Started | 34
Completed | 32
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 36 [20 to 75]
Age, Customized [Count of Participants; unit: Participants]
  20 - 30 years | 10
  31 - 40 years | 9
  41 - 60 years | 10
  61 - 75 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  More Than One Race | 1
  Other | 7
  White | 26
Region of Enrollment [Number; unit: participants]
  United States | 34
Stage [Count of Participants; unit: Participants] — Lugano Classification of disease stage
  * Stage I: Found in only 1 lymph node or lymphoid organ or the cancer is found in only 1 area of a single organ outside the lymph system.
  * Stage II: The cancer is found in 2 or more lymph node areas on the same side of the diaphragm or the cancer extends locally from one lymph node area into a nearby organ
  Can be assigned a letter A or B. B is when a patient has any of the following symptoms:
  * Loss of > than 10% of body weight over the previous 6 months without dieting
  * Unexplained fever of at least 100.4°F (38°C)
  * Drenching night sweats
  Participants
    IA | 6
    IIA | 24
    IIB | 4
Cellularity [Count of Participants; unit: Participants] — Hypercellular indicates more cells are being produce than expected, hypocellular means that fewer than expect number of cells are being produced, normocellular means an approximately normal amount of cells are being produced
  Participants
    Hypercellular | 1
    Hypocellular | 4
    Normocellular | 10
    Missing | 19
Histology [Count of Participants; unit: Participants] — The histological subtypes of classic Hodgkin lymphoma:
  * Classical NOS: Not Otherwise Specified (specific subtype not identified)
  * Lymphocyte-Rich: Rarely found in more than a few lymph nodes and usually occurs in the upper half of the body
  * Mixed Cellularity: Seen predominantly in adults, this is the second most common type. It can start in any lymph node but most often occurs in the upper half of the body.
  * Nodular Sclerosis: The most common type in developed countries. This most common in teens and young adults. Tends to start in lymph nodes in the chest or neck.
  Participants
    Classical Hodgkin Lymphoma, NOS | 8
    Lymphocytic Rich | 4
    Mixed Cellularity | 4
    Nodular Sclerosis | 18
Risk Class [Count of Participants; unit: Participants] — Early Unfavorable: Stage I or II disease and one or more of the following risk factors:
  * B Symptoms (see stage description)
  * Extranodal disease
  * Bulky disease (≥10 cm or >33% of the chest diameter on chest x-ray)
  * Three or more sites of nodal involvement
  * Sedimentation rate of ≥50 mm/h
  Early Favorable: Stage I or II disease with none of the risk factors listed above. Patients with favorable classification tend to have better outcomes.
  Participants
    Early Favorable | 21
    Early Unfavorable | 13
Number of Lesions [Median (Full Range); unit: Lesions] — Population: Information is missing for one participant
  Lesions
    number analyzed (Participants) | 33
    (all) | 5 [1 to 6]
Longest Tumor Diameter [Median (Full Range); unit: Centimeters (cm)] — Population: Information is missing for one participant
  Centimeters (cm)
    number analyzed (Participants) | 33
    (all) | 33.4 [15.1 to 83.3]

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Complete response rate at the end of therapy as measured by Positron emission tomography-computed tomography (PET/CT). Response is evaluated using Revised International Working Group Criteria. Complete response is defined as disappearance of all evidence of disease.
Time Frame: End of Therapy (median duration of four months)
Population: Two participants were not evaluated for response due to a death and a withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 32
Participants | 31

2. Secondary Outcome: Overall Response Rate After One Cycle of Brentuximab
Description: The number of participants achieving a Partial Response (PR) or Complete Response (CR) after one cycle of Brentuximab monotherapy as measured via PET/CT response. Response is evaluated using the Revised International Working Group Criteria.
  * CR: Disappearance of all evidence of disease
  * PR: Regression of measurable disease and no new sites
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
Participants | 18

3. Secondary Outcome: Overall Response Rate
Description: The number of participants achieving a Partial Response (PR) or Complete Response (CR) at the end of therapy as measured via PET/CT response. Response is evaluated using the Revised International Working Group Criteria.
  * CR: Disappearance of all evidence of disease
  * PR: Regression of measurable disease and no new sites
Time Frame: End of Therapy (median duration of four months)
Population: Two participants were not evaluated for response due to a death and a withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 32
Participants
  Complete Response | 31
  Partial Response | 0

4. Secondary Outcome: Grade III or IV Adverse Events
Description: A summary of the grade 3 or 4 adverse events experienced by participants as determined by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The data is shown as the number of participants that experienced at least one grade 3 or 4 adverse event for each of the specified toxicities.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
participants
  Peripheral sensory neuropathy | 8
  Neutrophil count decreased | 21
  Fatigue | 3
  Nausea | 1
  Anemia | 2
  White blood cell decreased | 6
  Abdominal pain | 2
  Diarrhea | 1
  Febrile neutropenia | 12
  Vomiting | 1
  Mucositis oral | 1
  Weight loss | 2
  Dehydration | 1
  Hypertension | 1
  Infections and infestations - Other, specify | 1
  Blood and lymphatic system disorders - Other, spec | 1

ADVERSE EVENTS:
Time Frame: From the start of therapy until the the end of followup due to disease progression, death, or withdrawal from the study. Median follow-up duration of 38 months.
Description: Adverse events were assessed with regularly scheduled physical exams, laboratory tests, and participant self reports.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/34
Serious Adverse Events (participants affected / at risk) | 15/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=34)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Neutrophil Count Decreased (Investigations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
White Blood Cell Decreased (Investigations) | 1 (2)
Viral Gastritis (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Bronchial Infection (Infections and infestations) | 1 (1)
Chest Pain - Cardiac (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1)
Hidradenitis Suppurativa (Skin and subcutaneous tissue disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Line Infection (Infections and infestations) | 1 (1)
Nausea, Vomiting, Dehydration (Gastrointestinal disorders) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 1 (1)
Anorexia, Fatigue (Metabolism and nutrition disorders) | 1 (1)
Hip pain, back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anorexia, Nausea, Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea, Hypotension (Gastrointestinal disorders) | 1 (1)
Fever, Sinus Congestion (General disorders) | 1 (1)
Ileus, Esophagitis, Transaminase elevation, low white blood cell count, dehydration (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=34)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 27 (52)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 3 (5)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 30 (53)
Fever (General disorders) | 4 (6)
Infusion related reaction (General disorders) | 3 (5)
Malaise (General disorders) | 2 (2)
Pain (General disorders) | 8 (14)
General disorders and administration site conditions - Other, (General disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (21)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 8 (12)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 14 (24)
Bloating (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 26 (35)
Diarrhea (Gastrointestinal disorders) | 15 (25)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (8)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 26 (41)
Oral pain (Gastrointestinal disorders) | 4 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 12 (18)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (8)
Upper respiratory infection (Infections and infestations) | 5 (7)
Urinary tract infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 4 (6)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 14 (21)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 10 (14)
Neutrophil count decreased (Investigations) | 26 (74)
Platelet count decreased (Investigations) | 6 (10)
Weight loss (Investigations) | 7 (14)
White blood cell decreased (Investigations) | 21 (56)
Investigations - Other, specify (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 5 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (17)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (21)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8)
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 9 (13)
Dizziness (Nervous system disorders) | 9 (9)
Headache (Nervous system disorders) | 9 (10)
Memory impairment (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 7 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 27 (67)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (5)
Anxiety (Psychiatric disorders) | 7 (8)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 12 (14)
Restlessness (Psychiatric disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 12 (31)
Hypotension (Vascular disorders) | 2 (3)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes